CLINICAL TRIAL: NCT05524181
Title: Telehealth-enabled Integrated Palliative Care for People With Dementia
Acronym: IBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Independence Blue Cross (Other)
Responsible Party: Principal Investigator, Brooke Worster, Principal Investigator, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 080-27000-U33701; #22G.239 (Other: Jefferson Institutional Review Board)
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Dementia of Alzheimer Type; Alzheimer Disease; Frontotemporal Degeneration; Lewy Body Dementia; Vascular Cognitive Impairment; Vascular Dementia; Mixed Dementia
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Dementia, Vascular; Mixed Dementias

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention or control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Individuals in the intervention group will undergo a series of two telehealth video visits and a series of survey assessments at baseline, 3, 6, 9, and 12 months.
  Interventions: Other: Telehealth Integrated Primary Care (TIPC)
- Control (No Intervention): Individuals in the control group will continue with their usual standard of care and undergo a series of survey assessments at baseline, 3, 6, 9 and 12 months.

INTERVENTIONS:
Other: Telehealth Integrated Primary Care (TIPC) — The TIPC model of intervention incorporates video visits across research clinicians and patients' existing care clinicians for more synergized and accessible care provision for a given clinical indication. The first TIPC visit will center around the patient setting care goals for themselves and their caregiver with the help of a palliative care physician. The second TIPC visit will focus on assessing goal attainment and also close the care loop between their existing care team, a research-appointed palliative care team, and their involvement in the study.
  Other Names: TIPC
  Arms: Intervention

SUMMARY:
In prior work, this team developed a telehealth primary care model (TIPC), designed in close partnership with patients and clinicians to address a widespread increase in telehealth use during the COVID-19 pandemic. This research team will test the TIPC intervention to assess support for patients among a population of persons with dementia (PwD). Participants will be enrolled in the study for a 12 month period.

This study's aims are 1) to explore the impact of the TIPC intervention on patient-important outcomes, engagement with community-based support provided through insurers, advanced care planning (primarily identification of health-care proxy), and patterns of hospice and healthcare utilization in the target population and 2) to evaluate patient, caregiver, and clinical team perspectives of feasibility and acceptability of a TIPC model, and apply findings from this work to the development of a larger randomized control trial designed to assess long-term efficacy of TIPC intervention.

DETAILED DESCRIPTION:
One in 3 deaths for those over the age of 65 are caused by Alzheimer's or related dementia. Lack of goals-of-care conversations with these patients drives up end-of-life healthcare costs due to excessive use of medical procedures and places unnecessary decision-making burden on caregivers. Such realities exhibit how existing models of specialty palliative care are suffering too great of a workforce shortage to adequately meet the needs of increasing numbers of PwD and are also inaccessible to underrepresented minorities (URMs) due to cost. Implementing a TIPC model could improve these outcomes through intersectional engagement of relevant health entities to carve more concrete care goals and drive down overall care cost.

This trial will enroll 50 patients and caregivers (when appropriate). Half of the patient participants will be given the TIPC intervention and all participants will be assessed over 12 months to assess changes in patient-important outcomes. For both groups, the researchers will evaluate goal attainment, quality of life, decision making, caregiver support/burden, and clinician/payor satisfaction. Assessments will be ongoing throughout the year (baseline, 3, 6, 9, and 12 months) to fully illustrate what kind of sustained impact or change in trajectory this brief intervention may have, and if other gaps are later identified.

Patient participants will be recruited from Jefferson EMR reports, physician referrals, and other forms of outreach. Patient participants will be randomly assigned to study groups (25 intervention, 25 control). If a patient is randomized to the intervention group, researchers will ask if they have a caregiver so that they may be enrolled in the study as well. Intervention subjects will partake in two telehealth visits as a part of the TIPC model. The first telehealth visit will focus on ACP and identifying patient-important outcomes via a web-based tool for discussion with a palliative care (PC) specialist. The second telehealth visit will involve patient communication of their patient important outcomes (PIOs) to a primary care provider (PCP) and the translation of those PIOs into care plans for ongoing management. Control subjects will be followed as they continue with their usual standard of care. They will also complete all measures at pre-specified time points and researchers will assess for changes in GAS, provider burden and decision making as well as hospitalizations, hospice, palliative care plans.

All patient/caregiver dyads assigned to the intervention group will be interviewed remotely after the intervention via survey to assess their goal attainment, satisfaction with care and connectivity to community resources.

Evaluation of patient outcomes of the TIPC model will be ongoing and through an assets/strengths-based framework. At baseline, 3, 6, 9, and 12 months, patient quality of life, decision-making, and caregiver support/burden will be measured through a series of follow-up assessments.

At 3, 6, 9, and 12 months, the degree to which intervention subjects felt each of their PIOs was met will be self-reported by the patient/caregiver.

To substantiate intervention impact on patients, both clinical and implementation outcomes (payor engagement, changes in level of care, recurrent hospitalizations, transition to hospice, intervention uptake, PCP satisfaction) will be measured and evaluated 6+ months post-intervention via retrospective data review. This is with the exception of PCP satisfaction which is to be self-reported following the same acceptability measures as the intervention subjects.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Individuals diagnosed with Alzheimer's Disease, Alzheimer's Disease Related Dementias, (including frontotemporal degeneration, Lewy body dementia, vascular contributions to cognitive impairment and dementia, or mixed etiology dementias), or patients billed for cognitive impairment in the last three years that have a Jefferson PCP
* Individuals with access to a smart phone, computer, or some other telehealth-capable technology
* English-speaking individuals

Exclusion Criteria:

* Traumatic Brain Injuries
* Incarceration
* Homelessness
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Change in Goal Attainment | 3 months
  Participants identify their own primary goals related to their care using the Goal Attainment Scaling (GAS) system, and report the degree to which each goal was met. Patients will set 2 concrete care goals and report if they feel like they met these goals much less than expected, less than expected, as expected, more than expected, or much more than expected.
Change in Goal Attainment | 6 months
  Participants identify their own primary goals related to their care using the Goal Attainment Scaling (GAS) system, and report the degree to which each goal was met. Patients will set 2 concrete care goals and report if they feel like they met these goals much less than expected, less than expected, as expected, more than expected, or much more than expected.
Change in Goal Attainment | 9 months
  Participants identify their own primary goals related to their care using the Goal Attainment Scaling (GAS) system, and report the degree to which each goal was met. Patients will set 2 concrete care goals and report if they feel like they met these goals much less than expected, less than expected, as expected, more than expected, or much more than expected.
Change in Goal Attainment | 12 months
  Participants identify their own primary goals related to their care using the Goal Attainment Scaling (GAS) system, and report the degree to which each goal was met. Patients will set 2 concrete care goals and report if they feel like they met these goals much less than expected, less than expected, as expected, more than expected, or much more than expected.
Change in Disease-Related Quality of Life | Baseline
  Participants report their overall quality of life by utilizing the Quality of Life in Alzheimer's Disease Scale (QoL-AD). These metrics include but are not limited to: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole. A summary index score is derived by applying an appropriate value set to the responses for each question (poor=1, fair=2, good=3, excellent=4). Patients can score up to 52 points with a higher score being associated with a higher quality of life.
Change in Disease-Related Quality of Life | 3 months
  Participants report their overall quality of life by utilizing the Quality of Life in Alzheimer's Disease Scale (QoL-AD). These metrics include but are not limited to: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole. A summary index score is derived by applying an appropriate value set to the responses for each question (poor=1, fair=2, good=3, excellent=4). Patients can score up to 52 points with a higher score being associated with a higher quality of life.
Change in Disease-Related Quality of Life | 6 months
  Participants report their overall quality of life by utilizing the Quality of Life in Alzheimer's Disease Scale (QoL-AD). These metrics include but are not limited to: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole. A summary index score is derived by applying an appropriate value set to the responses for each question (poor=1, fair=2, good=3, excellent=4). Patients can score up to 52 points with a higher score being associated with a higher quality of life.
Change in Disease-Related Quality of Life | 9 months
  Participants report their overall quality of life by utilizing the Quality of Life in Alzheimer's Disease Scale (QoL-AD). These metrics include but are not limited to: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole. A summary index score is derived by applying an appropriate value set to the responses for each question (poor=1, fair=2, good=3, excellent=4). Patients can score up to 52 points with a higher score being associated with a higher quality of life.
Change in Disease-Related Quality of Life | 12 months
  Participants report their overall quality of life by utilizing the Quality of Life in Alzheimer's Disease Scale (QoL-AD). These metrics include but are not limited to: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole. A summary index score is derived by applying an appropriate value set to the responses for each question (poor=1, fair=2, good=3, excellent=4). Participants can score up to 52 points with a higher score being positively associated with a higher quality of life.
Change in Decision-Making | Baseline
  Participants assess the extent to which they are involved in everyday decision making (e.g., when to get up, what foods to buy) the Decision-Making Involvement Scale (DMI). A summary index score is derived by applying an appropriate value set to the responses for each question (not at all involved=0, a little involved=1, fairly involved=2, very involved=3). Participants can score up to 45 points with a higher score being positively associated with a higher level of decision involvement.
Change in Decision-Making | 3 months
  Participants assess the extent to which they are involved in everyday decision making (e.g., when to get up, what foods to buy) the Decision-Making Involvement Scale (DMI). A summary index score is derived by applying an appropriate value set to the responses for each question (not at all involved=0, a little involved=1, fairly involved=2, very involved=3). Participants can score up to 45 points with a higher score being positively associated with a higher level of decision involvement.
Change in Decision-Making | 6 months
  Participants assess the extent to which they are involved in everyday decision making (e.g., when to get up, what foods to buy) the Decision-Making Involvement Scale (DMI). A summary index score is derived by applying an appropriate value set to the responses for each question (not at all involved=0, a little involved=1, fairly involved=2, very involved=3). Participants can score up to 45 points with a higher score being positively associated with a higher level of decision involvement.
Change in Decision-Making | 9 months
  Participants assess the extent to which they are involved in everyday decision making (e.g., when to get up, what foods to buy) the Decision-Making Involvement Scale (DMI). A summary index score is derived by applying an appropriate value set to the responses for each question (not at all involved=0, a little involved=1, fairly involved=2, very involved=3). Participants can score up to 45 points with a higher score being positively associated with a higher level of decision involvement.
Change in Decision-Making | 12 months
  Participants assess the extent to which they are involved in everyday decision making (e.g., when to get up, what foods to buy) the Decision-Making Involvement Scale (DMI). A summary index score is derived by applying an appropriate value set to the responses for each question (not at all involved=0, a little involved=1, fairly involved=2, very involved=3). Participants can score up to 45 points with a higher score being positively associated with a higher level of decision involvement.
Change in Caregiver Support/Burden | Baseline
  Caregivers of participants explore the personal and role strain that they experience via the Zarit Burden Inventory (ZBI22). A summary index score is derived by applying an appropriate value set to the responses for each question (never=1, rarely=2, sometimes=3, quite frequently=4, nearly always=5). Participants can score up to 88 points with a higher score being negatively associated with a higher level of burden experienced by the caregiver.
Change in Caregiver Support/Burden | 3 months
  Caregivers of participants explore the personal and role strain that they experience via the Zarit Burden Inventory (ZBI22). A summary index score is derived by applying an appropriate value set to the responses for each question (never=1, rarely=2, sometimes=3, quite frequently=4, nearly always=5). Participants can score up to 88 points with a higher score being negatively associated with a higher level of burden experienced by the caregiver.
Change in Caregiver Support/Burden | 6 months
  Caregivers of participants explore the personal and role strain that they experience via the Zarit Burden Inventory (ZBI22). A summary index score is derived by applying an appropriate value set to the responses for each question (never=1, rarely=2, sometimes=3, quite frequently=4, nearly always=5). Participants can score up to 88 points with a higher score being negatively associated with a higher level of burden experienced by the caregiver.
Change in Caregiver Support/Burden | 9 months
  Caregivers of participants explore the personal and role strain that they experience via the Zarit Burden Inventory (ZBI22). A summary index score is derived by applying an appropriate value set to the responses for each question (never=1, rarely=2, sometimes=3, quite frequently=4, nearly always=5). Participants can score up to 88 points with a higher score being negatively associated with a higher level of burden experienced by the caregiver.
Change in Caregiver Support/Burden | 12 months
  Caregivers of participants explore the personal and role strain that they experience via the Zarit Burden Inventory (ZBI22). A summary index score is derived by applying an appropriate value set to the responses for each question (never=1, rarely=2, sometimes=3, quite frequently=4, nearly always=5). Participants can score up to 88 points with a higher score being negatively associated with a higher level of burden experienced by the caregiver.

SECONDARY OUTCOMES:
Feasibility, Acceptability, and Satisfaction regarding TIPC Intervention | 3 months
  Participants in the intervention group will report their experience with the TIPC model via survey questions. Participants will indicate whether or not they strongly disagree, disagree, have no opinion, agree, or strongly agree with a series of statements asking them about their experience with TIPC intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05524181/ICF_000.pdf